CLINICAL TRIAL: NCT01862432
Title: Immediate Skin-to-skin Contact After Caesarean Delivery to Improve Neonatal
Brief Title: Immediate Skin-to-skin Contact After C-section
Acronym: CALIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Jean-Charles Pasquier, MD, PhD, Dr, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 10-097
Record Dates: First submitted 2013-05-15; First posted 2013-05-24 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Elective Cesarean Section; Term Birth (Pregnancy)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- immediate skin-to-skin (Experimental)
  Interventions: Other: Immediate skin-to-skin
- control (No Intervention)

INTERVENTIONS:
Other: Immediate skin-to-skin — The newborn is place on his mother's chest, immediately (in the first minute of life), in order to allow complete skin-to-skin contact.
  Arms: immediate skin-to-skin

SUMMARY:
At birth, the passage from intrauterine to the aerial life can be considered as one of the most stressful and painful life events. Skin-to-skin contact (STSC) with mother is known to provide numerous virtues and World Health Organisation (WHO) recently supported the introduction of such care among healthy, term-born neonates. Here, the investigators hypothesized that immediate STSC could reduce neonatal, birth-evoked stress and pain. This randomized controlled trial (RCT) aimed to compare the pain and stress response of C-section born neonates that received either immediate STSC with mother (intervention) or classical support and monitoring (control).

DETAILED DESCRIPTION:
Women are recruited before elective c-section.

Randomizatiion is performed just before the operation.

Control group:

The operation is performed as usual, with observation of the newborn by medical staff. The newborn is then wrapped in a blanket and given to the father.

Intervention group:

The newborn is given to the mother in the first minute of life, placed on her chest to allow complete skin-to-skin contact. Observation of the baby is performed in this position. The skin-to-skin contact lasts as long as the operation is not completed or the mother is not able anymore to keep her baby on her chest.

Sampling (in both groups):

* salivary samples are obtained with salivettes from the mother 1)before the operation and 2) after the operation, in the recovery room (90 minutes after birth).
* salivary samples are obtained with salivettes from the newborn 1) 20 minutes after birth and 2) 20 minutes after the vitamin K injection (performed at 60 minutes of life)
* A cord blood sample is obtained for prolactin, ACTH and cortisol analysis.

Video recording:

The newborn is video recorded at the vitamin K injection (from 1 minute before the injection to 5 minutes after) for analysis with the Neonatal Infant Pain Scale.

Satisfaction:

The mother's satisfaction is evaluated with a questionnaire 24 to 48 hours after birth.

Breastfeeding:

The breastfeeding is evaluated by a research nurse 1) at the hospital and 2) by phone interviews, up to 6 months after birth.

ELIGIBILITY:
Inclusion Criteria:

* elective C-section
* term pregnancy
* signature of an information and consent form

Exclusion Criteria:

* multiple pregnancy
* labor
* fetal distress
* abnormal anticipated birth weight
* congenital malformation
* diabetes
* fever
* rapid management of the new born required

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Breastfeeding at six months | six months

SECONDARY OUTCOMES:
Pain reactivity | one hour
  The newborn reactivity to pain is analyzed one hour after birth, at the injection of vitamin K, according to the Neonatal Infant Pain Scale.
mother's satisfaction | 48 hours
  Mother's satisfaction is evaluated by a questionnaire, within 48 hours after C-section.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles Pasquier, MD, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada